CLINICAL TRIAL: NCT02615509
Title: Comparison of the Philips MicroDose Tomosynthesis System to 2D Digital Mammography
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Discontinuation of development of device.
Sponsor: Philips Digital Mammography Sweden AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 9RWH8K
Record Dates: First submitted 2015-11-12; First posted 2015-11-26 (Estimated); Results first posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
Keywords: Mammography; Tomosynthesis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imaging on experimental tomo device (Other): Women will have a bilateral two-view mammogram (a total of four images) with the Philips MicroDose Tomosynthesis system and a bilateral two-view mammogram (a total of four images) with an FFDM system. The order of this will be randomised.
  After collecting the cases together with ground truth a readers study will be performed.
  Interventions: Radiation: Imaging on experimental tomo device

INTERVENTIONS:
Radiation: Imaging on experimental tomo device — The system used for imaging in the experimental arm is the Philips MicroDose tomography system. The system used for imaging in the active comparator is a standard FFDM system

SUMMARY:
The primary objective of this study is to compare the safety and clinical performance of the Philips MicroDose Tomosynthesis system images and images from FFDM systems.

DETAILED DESCRIPTION:
The study will be performed in two phases: Image Accrual and Image Reading.

Approximately 800 women who fulfill all inclusion and exclusion criteria will be enrolled in chronological order from up to 3 different US sites with one study investigator for each site. Two cohorts of patients will be enrolled (i.e., Biopsy and Screening Cohorts). Paired sets of a standard 4-view exam will be collected both from Philips Tomosynthesis system (Tomosynthesis and synthetic 2D images) and a FDA-cleared FFDM system. All enrolled cases will be quality controlled for completeness of image and patient information.

The reading portion of the study will include approximately 300 normal cases (including some cases determined to be normal after call back after screening mammography), 65 cancer cases, and 40 biopsy proven benign cases.

The primary objective of the study is to compare the safety and clinical performance of the Philips MicroDose Tomosynthesis system (Tomosynthesis and synthetic 2D) images to conventional 2D mammography images (FFDM).

ELIGIBILITY:
Inclusion Criteria:

* Patient is female and at least 40 years of age
* No contraindication for routine bilateral mammography

Screening Cohort

* Patient presents for a routine screening mammogram Biopsy Cohort
* Patient is scheduled for a biopsy
* Patient has a screening detected abnormality

Exclusion Criteria:

* Patient is pregnant or believes she may be pregnant; OR,
* Patient is breast feeding; OR
* Patient is unable or unwilling to give informed consent, including consent to reuse data for future research; OR,
* Patient has breast implants; OR
* Patient has previous surgical biopsy; OR
* Patient has previous breast cancer; OR
* Patient presented to screening with clinical symptoms (e.g. palpable lump, nipple discharge, nipple retraction, skin irritation or dimpling)

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2016-01; Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Etta Pisano, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with researchers outside the company or otherwise engaged in the study.

RESULTS

PARTICIPANT FLOW:
Groups:
- Imaging on Experimental Tomo Device: Women will have a bilateral two-view mammogram (a total of four images) with the Philips MicroDose Tomosynthesis system and a bilateral two-view mammogram (a total of four images) with an FFDM system. The order of this will be randomised.
  After collecting the cases together with ground truth a readers study will be performed.
  Imaging on experimental tomo device: The system used for imaging in the experimental arm is the Philips MicroDose tomography system. The system used for imaging in the active comparator is a standard FFDM system
Period: Overall Study
Arm/Group | Imaging on Experimental Tomo Device
Started | 347
Completed | 201
Not Completed | 146
Not completed — Lost to Follow-up | 134
Not completed — Death | 4
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Arm/Group | Imaging on Experimental Tomo Device
Number analyzed (Participants) | 347
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 243
  >=65 years | 104
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 347
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 347
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American indian or Alaskan native | 4
  Asian | 5
  African American | 105
  White | 233
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 347

OUTCOME MEASURES:

1. Primary Outcome: To Compare the Clinical Performance of the Philips MicroDose Tomosynthesis System Images to Conventional 2D Mammography Images. Clinical Performance Will be Based on the Area Under the Receiver Operating Characteristics Curve.
Description: Due to study termination the conventional images where not taken and it was not possible to calculate the Area under the Receiver Operating Characteristics Curve.
  Instead we are reporting the biopsy results from the Philips MicroDose Tomosynthesis system.
  The time frame from examination to biopsy is documented as an estimate based on the relative urgency to detect potential tumors.
Time Frame: Up to approximately 4 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Imaging on Experimental Tomo Device
Number analyzed (Participants) | 347
Participants
  Biopsy proven benign | 15
  Biopsy proven cancer | 14
  Negative recalled | 31
  Negative, no recall | 279
  Withdrawn | 8

2. Secondary Outcome: Compare Average Glandular Dose Between FDDM and Philips Tomosynthesis System
Time Frame: Nine months image accrual
Population: No data were collected due to study termination.
Arm/Group | Imaging on Experimental Tomo Device
Number analyzed (Participants) | 0

3. Secondary Outcome: Compare Non-cancer Recall Rates Between FDDM and Philips Tomosynthesis System.
Time Frame: Nine months image accrual
Population: No data were collected due to study termination.
Arm/Group | Imaging on Experimental Tomo Device
Number analyzed (Participants) | 0

4. Secondary Outcome: Compare Sensitivity Between FDDM and Philips Tomosynthesis System, Sensitivity Will be Estimated for Each Reader as the Proportion of Cancer Cases With Per-case BI-RADS Category 4 or Higher.
Time Frame: One year follow up will be performed on negative patients
Population: No data were collected due to study termination.
Arm/Group | Imaging on Experimental Tomo Device
Number analyzed (Participants) | 0

5. Secondary Outcome: Compare Specificity Between FDDM and Philips Tomosynthesis System. Specificity Will be Estimated by Reader as the Proportion of Non-cancer Cases With Per-case BI-RADS Category Less Than 4.
Time Frame: One year follow up will be performed on negative patients
Population: No data were collected due to study termination.
Arm/Group | Imaging on Experimental Tomo Device
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year.
Arm/Group | Imaging on Experimental Tomo Device
All-Cause Mortality (participants affected / at risk) | 4/347
Serious Adverse Events (participants affected / at risk) | 0/347
Other Adverse Events (participants affected / at risk) | 0/347

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT02615509/Prot_SAP_000.pdf